CLINICAL TRIAL: NCT05996575
Title: IMPACT: Investigating Mild Cognitive Impairment in Patients And Controls With TD-fNIRS
Brief Title: Investigating Mild Cognitive Impairment in Patients And Controls With TD-fNIRS
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: Kernel (Industry)
Responsible Party: Sponsor
Other Study IDs: KER2023-3-IMPACT
Record Dates: First submitted 2023-08-02; First posted 2023-08-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Mild Cognitive Impairment
Keywords: functional Near Infrared Spectroscopy (fNIRS); Aging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MCI Patients: Adult participants who are seeking neurological assessments for Mild Cognitive Impairment (MCI) at a participating clinic/study site.
  Interventions: Other: fNIRS measurement
- Healthy Controls: Healthy participants without a prior MCI or memory impairment diagnosis.
  Interventions: Other: fNIRS measurement

INTERVENTIONS:
Other: fNIRS measurement — Kernel Flow2 measurements.

SUMMARY:
The goal of the proposed observational, multi-site study is to use fNIRS neurophysiological data recorded during a battery of tasks to detect MCI within a cohort consisting of patients and age-matched healthy controls. Furthermore, the investigators aim to explore whether they can measure the severity of MCI symptoms in the patient population. If successful, this approach enables clinicians to track the disease at its source-the brain; possibly allowing for earlier detection of MCI and its progression, and ultimately more efficient interventions.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Must have a diagnosis of MCI (amnesiac or non-amnesiac) as determined by clinician
* Adults (older adults) between the ages of 55-85 years inclusive at time of enrollment
* Ability to perform informed consent on their own
* Fluent in English (speaking and reading)

Healthy Controls

* Adults (older adults) between the ages of 55-85 years inclusive at time of enrollment
* Ability to perform informed consent on their own
* Fluent in English (speaking and reading)

Exclusion Criteria:

Patients

* Alzheimer's or dementia diagnosis
* Current substance or alcohol dependence, and/or alcohol or substance abuse as determined by CAGE-AID assessment for drug and alcohol abuse. A score of 2 or higher would result in exclusion.
* Has uncorrected major visual or auditory deficits that would prevent them from completing a study task
* Current or recent (in the past 6 months) chemotherapy and/or radiation for any cancer
* Major medical illnesses and psychiatric conditions (other than MCI) including:

  * Severe/uncontrolled Diabetes, hypertension and hypothyroidism that could pose secondary causes of cognitive decline
  * Parkinson's disease
  * Motor neuron diseases
  * Multiple Sclerosis
  * Brain Tumor
  * Stroke
  * Encephalitis
  * Meningitis
  * Epilepsy
  * TBI with serious results (coma, unconscious for >2 hrs, or skull fracture)
  * Current serious psychiatric conditions (bipolar disorder, schizophrenia, or psychosis)

Healthy Controls

* Prior MCI or memory impairment diagnosis
* First-degree relative with dementia or clinically relevant memory problems
* Alzheimer's or dementia diagnosis
* Current substance or alcohol dependence, and/or alcohol or substance abuse as determined by CAGE-AID assessment for drug and alcohol abuse. A score of 2 or higher would result in exclusion.
* Has uncorrected major visual or auditory deficits that would prevent them from completing a study task
* Current or recent (in the past 6 months) chemotherapy and/or radiation for any cancer
* Major medical illnesses and psychiatric conditions including:

  * Severe/uncontrolled Diabetes, hypertension and hypothyroidism that could pose secondary causes of cognitive decline
  * Parkinson's disease
  * Motor neuron diseases
  * Multiple Sclerosis
  * Brain Tumor
  * Stroke
  * Encephalitis
  * Meningitis
  * Epilepsy
  * TBI with serious results (coma, unconscious for >2 hrs, or skull fracture)
  * Current serious psychiatric conditions (bipolar disorder, schizophrenia, or psychosis)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult participants seeking neurological assessments for Mild Cognitive Impairment (MCI) at a participating clinic/study site. A separate cohort of age-matched healthy participants will be recruited as the control group. The current study, including the acquired data and participation in the study, has no influence on diagnosis or treatment decisions.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Brain hemodynamic activity with TD-fNIRS | About 1 hour during the study visit
  This includes changes in the concentration of oxygenated and deoxygenated hemoglobin as measured by the change in light absorption.
Optical properties of the brain with TD-fNIRS | About 1 hour during the study visit
  This measures how much light is absorbed at different points on the head.
Physiological features with TD-fNIRS | About 1 hour during the study visit
  This includes cardiac measures, such as heart rate (HR) and heart rate variability (HRV).

SECONDARY OUTCOMES:
Mini-Mental State Evaluation (MMSE) | Within 6 months of the study visit
  Clinician-administered screening tool used to systematically and thoroughly assess mental status through five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. Patient cohort only. Scores range between 0-30. A score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be abnormal, indicating possible cognitive impairment.
Mini-Cog | About 30 minutes during the study visit
  A fast and simple screening test to help detect cognitive impairment in its early stages that will be used to confirm normal cognitive function in the control group. Healthy control cohort only. Scores range between 0-5. Participants who score 0-2 are considered to indicate higher likelihood of cognitive impairment.
Geriatric Depression Scale (Short Form) | About 30 minutes during the study visit
  15-item self report measure of depression in older adults. Scores range between 0-15. Higher scores indicate high severity of depression.
General Anxiety Disorder | About 30 minutes during the study visit
  Seven-item self report measure used to assess participant anxiety. Scores range between 0-21. Higher scores indicate high severity of anxiety.
Apathy Evaluation Scale | About 30 minutes during the study visit
  18-item self-rated measure used to assess and quantify emotional, behavioral, and cognitive aspects of apathy. Scores range between 18-72. Higher scores indicate high severity of apathy.
Alzheimer's Disease Cooperative Study Activities of Daily Living for Mild Cognitive Impairment (ADCS ADL-MCI) | About 30 minutes during the study visit
  15-item self report measure used to assess performance of activities of daily life. Scores range between 0-45. Higher scores indicate declining cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Perdue, PhD, Principal Investigator — Kernel
Locations (6):
- United States (6):
  - The Research Center of Southern California, Carlsbad, California
  - BrainHealth Solutions, Costa Mesa, California
  - The Research Center of Southern California, Escondido, California
  - Kernel, Los Angeles, California
  - Syrentis Clinical Research, Santa Ana, California
  - The Research Center of Southern California, Temecula, California

IPD SHARING:
Plan to Share IPD: Undecided